CLINICAL TRIAL: NCT01279902
Title: Phase 2 Study of Abbreviated 3 Cycles of Rituximab Plus CHOP (Cyclophosphamide, Adriamycin, Vincristine, and Prednisolone) Immunochemotherapy in Patients With Completely Excised Stage I or II CD20+ Diffuse Large B-cell Lymphoma
Brief Title: Abbreviated R-CHOP in Completely Excised Stage I or II DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Cheolwon Suh, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC_NHL01
Record Dates: First submitted 2010-08-03; First posted 2011-01-20 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large B-cell lymphoma; rituximab; CHOP; abbreviated therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab plus CHOP Immunochemotherapy (Experimental): Interventions: conventional R-CHOP every 3 weeks for 3 cycles
  * Rituximab 375 mg/M2 IV day 1
  * Cyclophosphamide 750 mg/M2 IV day1
  * Vincristine 1.5 mg/M2 (max. 2 mg) IV day1
  * Prednisolone 50 mg bid day 1-5, every 3 weeks
  Interventions: Drug: Rituximab plus CHOP Immunochemotherapy

INTERVENTIONS:
Drug: Rituximab plus CHOP Immunochemotherapy — The R-CHOP treatment will continue up to 3 cycles with interval of 21 days: Each cycle consists of rituximab 375mg/m2 (iv, on day 1), cyclophosphamide 750 mg/m2 (iv, on day 1), doxorubicin 50mg/m2 (iv, on day 1), vincristine 1.4mg/m2 (iv, on day 1), and prednisolone 100mg (po, on day 1-5).

SUMMARY:
This study aims; to assess the efficacy of shortened systemic chemotherapy in patients with completely excised CD20 positive Diffuse Large B-cell Lymphoma (DLBCL) with Ann Arbor Stage I or II.

DETAILED DESCRIPTION:
Unlike the limited stage diffuse Large B-cell Lymphoma (DLBCL) treated with primary chemotherapy followed by radiotherapy, patients with stage I or II DLBCL would be treated with surgical resection followed by chemotherapy in this trial. While chemotherapy is the main treatment modality and radiotherapy becomes adjuvant treatment in the former treatment scheme, surgical resection will remove all the gross lesions and chemotherapy aims to remove all microscopic disease whichever exists in the latter treatment scheme. Currently, six cycles of chemotherapy is usually performed after surgery even without any residual lesion compared with three cycles of chemotherapy in the former treatment scheme which plays primary role in the treatment scheme. The investigators will investigate whether abbreviated 3 cycles of Rituximab Plus Cyclophosphamide, Adriamycin, Vincristine, and Prednisolone (R-CHOP) immunochemotherapy following complete resection is an effective and safe treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent curative resection of primary tumor
* Pathologically confirmed CD20 positive diffuse large B-cell lymphoma (DLBCL) after surgical resection
* Ann Arbor Stage I or II
* No history of chemotherapy
* Performance status: ECOG 0-2
* Age: 18 to 70 years old
* Complete excision with negative resection margin on pathologic report after surgery
* Cardiac ejection fraction ≥ 50% as measured by MUGA or 2D echocardiography without clinically significant abnormalities
* Adequate renal function: serum creatinine level below 2 mg/dL (177μmol/L)
* Adequate liver functions: Transaminase (AST/ALT) < 3X upper normal value, Bilirubin < 2X upper normal value
* Adequate hematologic function: hemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1,500/mm3 and platelet count ≥ 75,000/mm3
* Informed consent

Exclusion Criteria:

* Patients with a known history of HIV (+) or HCV (+). However, HBV(+) patients are eligible if primary prophylaxis is given
* Previous or concurrent cancer that is distinct in primary site or histology from DLBCL, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions

  1. Unstable cardiac disease (i.e. congestive heart failure, arrhythmia symptomatic coronary artery disease) despite treatment, myocardial infarction within 6 months prior to study entry
  2. History of significant neurological or psychiatric disorders including dementia or seizures
  3. Active uncontrolled infection (viral, bacterial or fungal infection)
  4. Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or their ingredients
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy
* Patient with B symptoms or Bulky disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  Proportion of patients surviving 2 years after first R-CHOP chemotherapy with no relapse of DLBCL

SECONDARY OUTCOMES:
Overall survival | 2 years
  proportion of patients surviving at 2 year after first cycle of R-CHOP chemotherapy regardless of relapse of DLBCL
any adverse events as a measure of safety and tolerability | from the first R-CHOP to 1 month after completion of R-CHOP
  The number of patients with adverse events will be measured during R-CHOP chemotherapy according to CTCAE version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, MD, PhD, Principal Investigator — Asan Mecical Center, University of Ulsan College of Medicine
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang S, Cho H, Sohn BS, Oh SY, Lee WS, Lee SM, Yang DH, Huh J, Yoon DH, Suh C. Long-term follow-up of abbreviated R-CHOP chemoimmunotherapy for completely resected limited-stage diffuse large B cell lymphoma (CISL 12-09). Ann Hematol. 2020 Dec;99(12):2831-2836. doi: 10.1007/s00277-020-04284-z. Epub 2020 Sep 28. PMID 32989495